CLINICAL TRIAL: NCT02687698
Title: Effect of a Lipidic and Proteic Controlled Diet on Resting Energy Expenditure, Body Composition and Symptoms in Patients With Parkinson's Disease
Brief Title: Effect of a Lipidic and Proteic Controlled Diet on Parkinson's Disease
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: University of Padova (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 3575/AO/15
Record Dates: First submitted 2016-02-08; First posted 2016-02-22 (Estimated); Last update posted 2016-02-22 (Estimated); Status verified 2016-02

CONDITIONS: Parkinson Disease
MeSH Terms: conditions — Parkinson Disease | interventions — Diet, Ketogenic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Ketogenic diet (Experimental): Patients will be suggested to follow a ketogenic diet for 8 weeks.
  Interventions: Other: Ketogenic diet
- Control (No Intervention): Usual diet.

INTERVENTIONS:
Other: Ketogenic diet — The proposed ketogenic diet will concern a low glucidic diet with 60-70% of lipidic intake and 20-30% of proteins.
  Arms: Ketogenic diet

SUMMARY:
Parkinson's disease concerns some defects in carbohydrates metabolism involved in the progress of the pathology. Ketogenic diet has been largely studied as treatment on drug-resistant epilepsy and other neurologic diseases, but there is little information on the impact of this kind of diet in clinical aspects of Parkinson's disease. The aim of our study is thus to evaluate the effect of a lipid and protein controlled diet on resting energy expenditure, body composition and symptoms in patients with Parkinson's disease.

DETAILED DESCRIPTION:
Parkinson's disease concerns some defects in carbohydrates metabolism involved in the progress of the pathology. Ketogenic diet has been largely studied as treatment on drug-resistant epilepsy and other neurologic diseases, but there is little information on the impact of this kind of diet in clinical aspects of Parkinson's disease. The aim of our study is thus to evaluate the effect of a lipid and protein controlled diet on resting energy expenditure, body composition and symptoms in Parkinson's disease patients.

ELIGIBILITY:
Inclusion Criteria:

* patients with a diagnosis of Parkinson's disease, treated with L-Dopa or other dopaminergic drugs.
* Mini Mental State Examination (MMSE) >24.
* Activities of Daily Living >3.

Exclusion Criteria:

* Mini nutritional assessment <17; BMI <18, hypoalbuminemia or lymphopenia.
* acute or chronic liver diseases;
* renal function impairment (Clearance creatinine <30ml/min);
* cancer;
* acute inflammatory diseases;
* thyroid diseases;
* diabetes mellitus;
* dysphagia;
* dementia;
* dyslipidemia;
* history of recent cardiovascular or cerebrovascular events;
* psychiatric diseases;
* iatrogen parkinsonism.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2016-02; Primary Completion 2017-02 (Estimated); Study Completion 2017-02 (Estimated)

PRIMARY OUTCOMES:
Changes in resting energy expenditure | Baseline, week 4 and week 8
  Changes in resting energy expenditure as measured by indirect calorimetry

CONTACTS AND LOCATIONS:
Overall Officials: Caterina Trevisan, MD, Principal Investigator — University of Padova, Geriatric Section
Locations (1):
- Geriatric Section, Padua, Padova, Italy

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Vanitallie TB, Nonas C, Di Rocco A, Boyar K, Hyams K, Heymsfield SB. Treatment of Parkinson disease with diet-induced hyperketonemia: a feasibility study. Neurology. 2005 Feb 22;64(4):728-30. doi: 10.1212/01.WNL.0000152046.11390.45. PMID 15728303
- [Derived] Shehu E, Trevisan C, Sambo S, Ceolin C, Pavan S, Piazzani F, Sergi G, March A. Sex Differences in the Burden of Hip Fractures on Functional Status in Older Age. J Womens Health (Larchmt). 2023 Jan;32(1):57-62. doi: 10.1089/jwh.2021.0270. Epub 2022 Dec 1. PMID 36459629